CLINICAL TRIAL: NCT03797066
Title: Localized on -Site Testing and Treatment of Hepatitis C in Homeless Persons in South London: a Pilot Non-randomised Phase 4 Interventional Clinical Trial of Grazoprevir and Elbasvir ± Ribavirin in Participants With Genotype 1a, 1b or 4 to Measure Efficacy and Adherence to Treatment in a Homeless Population
Brief Title: ATTIC - Access To Treat in the Community
Acronym: ATTIC
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Changing parameters in HCV management, resulted in poor recruitment; additionally onset of SARS CoV2 resulted in the cessation of all mobile clinical services.
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Hepatitis C Trust (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KCHATTIC01
Record Dates: First submitted 2018-10-30; First posted 2019-01-08 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Hepatitis C, Chronic
Keywords: hepatitis C virus; homeless
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — elbasvir-grazoprevir drug combination

STUDY DESIGN:
Intervention Model Description: non-randomised, open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single arm (Other): A phase 4, open label, non-randomised study, conducted in hostels and homeless shelters in London; as well as mobile clinics in collaboration with the Hep C trust and the NHS Find and Treat program.
  Treatment: 12 or 16 weeks of Zepatier, based on genotypes; with Ribavarin for certain subtypes. The study drug is administered as a single tablet; which is a combination of 100 mg of grazoprevir and 50 mg of elbasvir; as outlined below:
  Genotypes 1a/b and 4: once daily dose for 12 weeks, taken with / without food. Genotype 1a and 4: (HCV RNA> 800,000 iu/ml or baseline NS5A resistance): once daily dose for 16 weeks, taken with / without food.
  NO dose modifications with the study drug.
  Interventions: Drug: ZEPATIER 50Mg-100Mg Tablet

INTERVENTIONS:
Drug: ZEPATIER 50Mg-100Mg Tablet — Zepatier 50/100 OD , with addition of Ribavarin in patients with Genotype 1a and 4 with HCV RNA> 800,000 iu/ml or baseline NS5A resistance.

SUMMARY:
The study is looking at the potential of utilizing a "point of care" test and treat pathway; using the DDA called Zepatier for achieving SVR in an homeless population who have tested positive for genotype 1 or 4 HCV.

DETAILED DESCRIPTION:
Direct acting antivirals (DAA) are new medications that have been approved for the management of HCV. These drugs have proven to be very effective in curing the HCV, without the need for interferon injections; which have always been used in the past. There are many combinations of DAAs, which treat specific types of HCV. Persons who test positive for the virus are typically referred to be seen and treated by a specialist hepatitis service based in hospital. This means that individuals may sometimes not attend the hospital to commence treatment; or follow up on their management.

The study is designed to explore if testing and treating individuals close to their own "local" setting will be an improvement to the current treatment pathway and encourage better involvement with the health care team; as well as looking at what the health care team can do to ensure participants in this test-and-treat trial receive the entire course of drug treatment prescribed to treat their HCV infection.

Participants infected with either genotype 1 or 4 HCV infection will be treated with Zepatier, a DAA which works by stopping the hepatitis C virus from (multiplying). The study medication is taken for 12 or 16 weeks depending on the genotype (or strain of HCV). Some participants will be given an additional drug called ribavirin. The study will examine the effectiveness of Zepatier at clearing the hepatitis C virus from the blood and body; and also what particular effects may be experienced by participants who may also be taking treatment for other conditions. Participants affected with other genotypes (not 1 and 4)will be offered standard NHS treatment with the appropriate antiviral combination for these strains.

ELIGIBILITY:
Inclusion Criteria:

1. Participants 18 years or older with chronic hepatitis C genotype 1 or 4 will be eligible.
2. Able and wiling to provide written informed consent.
3. Both interferon treatment naïve and experienced participants will be included.
4. Participants without cirrhosis will be eligible if HCV RNA positive, documented chronic hepatitis C and a FibroScan of ≤ 12.5.
5. Participants with cirrhosis (Fibroscan > 12.5 or APRI > 2) will be eligible if the serum albumin is > 3.5 g/dl, platelets > 100,000 and INR < 1.5 and there is no prior history of hepatic decompensation.
6. Participants with well controlled HIV coinfection will be included, but should be stabilized on antiretrovirals for which no clinically significant interaction is expected.
7. Participants who are HBsAg positive will be included, but will require antiviral prophylaxis for HepB. Anti- HbC positive participants will be included. Prophylaxis will not be given, but these participants will require careful monitoring of their ALT levels.

Exclusion Criteria:

* Persons with prior HCV DAA treatment
* Individuals younger than 18 years of age
* Individuals infected with genotypes other than 1a or 1b or 4 HCV identified on screening; however such participants identified on screening will be offered appropriate NHS England standard of treatment for the genotype.
* Unable or unwilling to give informed consent
* Active tuberculosis
* Females who are pregnant, planning pregnancy or breastfeeding
* Concurrent and/or recent involvement in other research that is likely to interfere with the intervention within three months of study enrolment
* Clinically-significant medical or psychiatric illness (other than chronic HCV) in the past, present, or being evaluated, that may interfere with participant treatment, safety, assessment or compliance with the protocol
* Participants with cirrhosis (Fibroscan > 12.5 or APRI > 2) and serum albumin is < 3.5 g/dl, platelets <100,000 and INR > 1.5 or a prior history of hepatic decompensation
* Severe renal impairment with eGFR <30 mL/min/1.73m2 or requiring dialysis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-03-23 (Actual); Primary Completion 2020-07-28 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
SVR | 24 months
  The percentage of participants achieving an SVR, defined as an HCV RNA evel less than the lower limit of quantification by sensitive PCR; by means of a short directed test and treat program in the homeless community.

SECONDARY OUTCOMES:
prevalence of HCV infection | 24 months
  Reduction in local prevalence of of viraemic hepatitis C, after a pilot trial of treatment in three to four homeless hostels.
Baseline knowledge evaluation | 24 months
  Participant knowledge of their hepatitis C status (disease, diagnosis, and current available approved treatments) will be assessed by means of a questionnaire completed at baseline. The researchers will also review participants willingness to engage in a test and treat protocol and correlate these findings with demographic and sociological data. This will be done using a questionnaire designed by the researchers; containing simple questions with respect to currently available testing and treatment of HCV infection.
Change From Baseline (BL) to SVR12 timepoint in 36-Item Short-Form Health Survey (SF-36) Scores | baseline, SVR 12 (twelve weeks post end of active treatment/ last dose of study drug)
  The 36-Item Short Form Health Survey (SF-36) is a set of generic, coherent, and easily administered quality-of-life measures. The survey addresses eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health. Participants self-report on items in a subscale that have between 2-6 choices per item using Likert-type responses (e.g. none of the time, some of the time, etc.). Summations of item scores of the same subscale give the subscale scores, which are transformed into a range from 0 to 100; zero= worst HRQL, 100=best HRQL.
  Data will be analysed ffg the guidelines suggested by the developers https://www.rand.org/health/surveys_tools/mos/36-item-short-form/scoring.html
Change From Baseline (BL) to SVR 12 in Chronic Liver Disease Questionnaire-Hepatitis C Virus (CLDQ-HCV) | baseline , SVR 12 (twelve weeks post end of active treatment/last dose of study drug)
  Impact of a localized test and treat protocol on health related quality of life will be assessed using the CLDQ-HCV instruments. The CLDQ-HCV is a disease-specific questionnaire measuring HRQL that contains 29 items divided into 4 domains: emotional function (9 items), worry (6 items), systemic symptoms (8 items) and activity/energy (6 items). All items refer to the previous 2 weeks and are rated on a 7 point Likert scale, with 1 corresponding to the maximum frequency ("all of the time") and 7 to the minimum ("none of the time"). Domain scores are the means of the items contained. A summary score is calculated by the mean of all domain scores (CLDQ-HCV Global). Higher scores indicate better health-related quality of life
Percentage of Participants Who Were Compliant With Treatment According To Moriskey, Green And Levine Adherence Scale (MAS4)(Subset Analysis) | 12 or 16 weeks
  Adherence to treatment measured by Moriskey, Green and Levine Adherence scale. This is a 4 item questionnaire that is easy to administer and score (using a yes/no format); and quickly identifies barriers to adherence.An answer of yes to zero questions indicates high adherence behavior, answering yes to one or two questions indicates medium adherence behavior, and answering yes to three or four questions indicates low adherence behavior
Percentage of Participants Who Were Compliant With Treatment According To Medication Count (Subset Analysis) | 12 or 16 weeks
  Compliance will be calculated as the amount of dispensed medication minus the amount of medication returned by participants at each visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Kings College Hospital NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
anonymised data sharing only, via publications